CLINICAL TRIAL: NCT00604552
Title: AneuRx Post Market Surveillance Registry
Brief Title: AneuRx Post Market Study in the Treatment of AAA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Mutual agreement between FDA closed the 522 postmarket surveillance Registry.
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS01000010
Record Dates: First submitted 2007-12-21; First posted 2008-01-30 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aneurysm
Keywords: Abdominal Aneurysm; Endovascular Aortic Repair (EVAR); Endovascular Stent Graft; Endograft
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifeline Registry (Other): All comers registry for the on-label treatment of AAA with the AneuRx Stent Graft sponsored by the Foundation of Society for the Vascular Surgery (SVS)
  Interventions: Device: AneuRx Stent Graft
- PS Registry (Other): All comers registry for the on-label treatment of AAA with the AneuRx Stent Graft sponsored by Medtronic
  Interventions: Device: AneuRx Stent Graft

INTERVENTIONS:
Device: AneuRx Stent Graft — Abdominal Aortic Aneurysm Repair

SUMMARY:
The aorta is a large blood vessel that carries blood away from the heart to the organs in the rest of the body. An aneurysm is a weakening in the artery wall that will become a bulge in the aorta. If left untreated, this bulge may continue to grow larger and may rupture (break open) with fatal consequences. Abdominal aortic aneurysm (AAA) is a life-threatening lesion that has been treated in recent year via endovascular repair.

The purpose of this study is to monitor the long term performance of the AneuRx Stent Graft Systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with an AneuRx Stent Graft per Instructions for Use
* Patients must provide written informed consent and agree to be accessible for follow-up at the study center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2003-07; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medtronic Cardiovascular, Study Chair — Medtronic
Locations (8):
- United States (8):
  - Tucson, Arizona
  - Royal Oak, Michigan
  - Morristown, New Jersey
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifeline Registry | PS Registry
Started | 189 | 160
Completed | 189 | 160
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifeline Registry | PS Registry | Total
Number analyzed (Participants) | 189 | 160 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (8.53) | 74.3 (7.31) | 75.1 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 21 | 51
  Male | 159 | 139 | 298
Region of Enrollment [Number; unit: participants]
  United States | 189 | 160 | 349

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Occurrence of Death, Aneurysm Rupture, and Surgical Conversion
Description: Number of patients that had an occurrence of death, aneurysm rupture or surgical conversion
Time Frame: 5 year
Population: All those treated on-label for the treatment of an AAA and followed out to 5 years.
Measure: Number; unit: participants
Arm/Group | Lifeline Registry | PS Registry
Number analyzed (Participants) | 189 | 160
participants
  Death | 21 | 20
  Aneurysm Rupture | 0 | 1
  Surgical Conversion | 1 | 2

2. Secondary Outcome: Evaluate the Occurance of Endoleak, Stent Graft Migration, Aneurysm Enlargement, Device Integrity and Adverse Events
Time Frame: 5 years
Population: Study terminated before subjects met study 5 year endpoints. FDA agreed to closure of study prior to reaching the 5 year endpoint.
Arm/Group | Lifeline Registry | PS Registry
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Lifeline Registry | PS Registry
Serious Adverse Events (participants affected / at risk) | 0/189 | 0/160
Other Adverse Events (participants affected / at risk) | 0/189 | 0/160

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No